CLINICAL TRIAL: NCT02912143
Title: German Pediatric Hemophilia Research Database
Acronym: GEPHARD
Status: Recruiting | Type: Observational
Sponsor: Goethe University (Other)
Collaborators: Society for Thrombosis and Haemostasis Research (Germany) (Other)
Responsible Party: Principal Investigator, Christoph Königs, Consultant Pediatric Hemophilia Center, Goethe University
Other Study IDs: GEPHARD; DRKS00011101 (Registry Identifier: DRKS)
Record Dates: First submitted 2016-09-17; First posted 2016-09-23 (Estimated); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Hemophilia A; Hemophilia B; Children; Drug Specific Antibodies
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- newly diagnosed children with hemophilia: no intervention
  Interventions: Other: documentation only

INTERVENTIONS:
Other: documentation only

SUMMARY:
The German Pediatric Hemophilia Research Database will collect data on the prophylactic and therapeutic use of factor concentrates, complications, outcome measures (joint scores, QoL) and living circumstances in newly diagnosed children with hemophilia.

ELIGIBILITY:
Inclusion Criteria:

* hemophilia A or B
* FVIII/FIX <1% to 25%
* informed consent

Exclusion Criteria:

* no consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children between 0 and 18 yrs diagnosed with hemophilia A or B (FVIII/FIX < 1% to 25%) from 01.01.2017.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-01-01; Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with antibody developement to exogenous clotting factors (>0.5 BU) | 5 years
  Blood Test: measurement in Bethesda Units, positive according to local standards, for most labs > 0.5 BU

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Königs, PhD, Principal Investigator — Goethe University
Locations (1):
- Goethe University, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No
Individual Patient data will not be shared outside specified collaborating studies (none yet)